CLINICAL TRIAL: NCT03138772
Title: Tracking CF Lung Disease Through the Early Years: Utility of the LCI
Acronym: LCITRACK
Status: Completed | Type: Observational
Sponsor: Felix Ratjen (Other)
Responsible Party: Sponsor-Investigator, Felix Ratjen, Principal Investigator, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 1000055762
Record Dates: First submitted 2017-04-27; First posted 2017-05-03 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Observational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: No intervention. Only monitoring LCI
  Interventions: Other: This is an observational study, no intervention used.
- Cystic Fibrosis Patients: No intervention. Only monitoring LCI
  Interventions: Other: This is an observational study, no intervention used.

INTERVENTIONS:
Other: This is an observational study, no intervention used. — No intervention is being used in this study.

SUMMARY:
This is a prospective observational study to follow a cohort of patients with Cystic Fibrosis and healthy controls for a period of two years. This study will include monitoring the subjects lung clearance index (by performing a breathing test called the multiple breath washout), as well as spirometry and their respiratory symptoms every three months as well as during a pulmonary exacerbation and after their recovery.

DETAILED DESCRIPTION:
This is a prospective observational cohort study. During the 3 year study period, each participant will be followed for a period of 2 years. The study will include quarterly measurements of the lung clearance index (LCI), as well as spirometry, for CF patients at their routine clinic visits. Parents of patients with CF will be asked to call the study nurse or clinical nurse if they experience a worsening of pulmonary symptoms and to come to the clinic for assessment of lung function. CF patients will then be assessed by a CF physician to assess whether they require antibiotic treatment based on a clinicians decisions to treat with antibiotics. The treatment decision will be left to the discretion of the patient's responsible physician, who will be blinded to the MBW results. All patients who meet the symptom based definition of a pulmonary exacerbation, regardless of treatment decision, will have MBW measured after 4 weeks. Following these visits at the time of an exacerbation, patients will have their MBW measured at their next clinic visit (usually within 3 months), and every 3 months thereafter until the end of the 2 year observation period, or the repeat onset of symptoms.This study will capture a maximum of two exacerbations per patient over the 2 year study period.

ELIGIBILITY:
Inclusion Criteria for Healthy Controls:

* Informed consent by patient or parent/legal guardian, verbal assent where appropriate
* Age 3 years to 16 years old
* Clinically stable with no signs of an acute exacerbation at enrollment visit
* Previously participated in a longitudinal MBW study at the Hospital for Sick Children and at the Riley Hospital for Children

Inclusion Criteria for CF Patients:

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent by patient or parent/legal guardian, verbal assent where appropriate
* Age 3 years to 16 years old
* Clinically stable with no signs of an acute exacerbation at enrollment visit

Exclusion Criteria:

* Previous organ transplantation
* Chronic lung disease not related to CF, such as asthma
* Use of intravenous antibiotics or other course of oral antibiotics (excluding maintenance treatment antibiotics) within 14 days of enrollment visit
* Physical findings at screening that would compromise the safety of the participant or the quality of the study data

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: There were 139 subjects recruited in the original preschool longitudinal study, and all participants from this original study will be invited to participate in this follow up study. We would like to recruit an additional 40 CF patients at the Hospital for Sick Children to increase our cohort size.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Lung Clearance Index | an average of 2 years
  Outcome measure from the Multiple Breath Washout test.

SECONDARY OUTCOMES:
Spirometry | an average of 2 years
  FEV1
Respiratory Cultures | an average of 2 years
  Bacterial pathogens IL-8 and neutrophil elastase
Respiratory Symptoms | an average of 2 years
  CFQ-R
Respiratory Symptoms | an average of 2 years
  CFRSD-CRISS

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No